CLINICAL TRIAL: NCT06908616
Title: The Prevalence of Ethnic Neutropenia in Neonates
Brief Title: Prevalence of Ethnic Neutropenia and Duffy Null Phenotype in Neonates
Status: Recruiting | Type: Observational
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Tal Ben-Ami, Head of Pediatric Hemato-Oncology, Kaplan Medical Center
Other Study IDs: KMC-24-0090; KMC-24-0090 (Other: Kaplan Medical Center Ethical Committee)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neutropenia (Low White Blood Cell Count)
Keywords: Neonates; Neutropenia; Duffy null associated count
MeSH Terms: conditions — Neutropenia; Leukopenia | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonatal birth cohort: Neonates born at Kaplan Medical Center whose cord blood is tested for Duffy antigen status and complete blood count. Follow-up neutrophil data is collected at 9-12 months if available.
  Interventions: Diagnostic Test: Cord blood

INTERVENTIONS:
Diagnostic Test: Cord blood — Cord blood samples will be collected during routine G6PD testing. An additional 3 mL will be obtained non-invasively from the umbilical cord to determine the expression of Duffy antigens using serologic gel testing.

SUMMARY:
This is a prospective observational study designed to assess the prevalence of the Duffy null phenotype (associated with ethnic neutropenia) in neonates born at Kaplan Medical Center. Blood samples will be collected from umbilical cords (non-invasively) to evaluate Duffy antigen expression. Data on ethnicity, perinatal factors, and routine blood counts at 9-12 months (when available) will also be collected to correlate phenotype with absolute neutrophil count (ANC).

DETAILED DESCRIPTION:
This is a prospective, observational cohort study designed to evaluate the prevalence of the Duffy null phenotype (Fya-/Fyb-) and its association with ethnic neutropenia in neonates born at Kaplan Medical Center in Israel. The Duffy null phenotype has been linked to lower peripheral neutrophil counts without increased infection risk in certain ethnic groups, a condition commonly referred to as benign ethnic neutropenia.

Cord blood samples will be collected from approximately 1,000 neonates during routine G6PD testing. An additional 3 mL will be obtained non-invasively from the umbilical cord after labour to determine the expression of Duffy antigens using serologic gel testing. Parental consent will be obtained, and information regarding ethnicity and family history of neutropenia will be collected.

Participants identified with the Duffy null phenotype will be followed through electronic health records to assess their neutrophil counts during routine blood screening at 9-12 months of age. The study will analyze associations between Duffy phenotype, neutropenia prevalence, and parental ethnic origin.

Findings may support improved diagnostic clarity around neonatal neutropenia and help reduce unnecessary interventions in otherwise healthy infants with genetically determined low neutrophil counts.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at Kaplan Medical Center between 1.9.2024 and 31.12.2025
* Parental informed consent obtained
* Umbilical cord blood available for routine testing

Exclusion Criteria:

* None

Ages: 1 Minute to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates born at Kaplan Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Duffy null phenotype in neonates | At birth (umbilical cord sample)
  Percentage of neonates born with the Duffy null phenotype (Fya-/Fyb-) as determined by serologic gel-based testing.

SECONDARY OUTCOMES:
Prevalence of neutropenia in infants with Duffy null phenotype | 9-12 months
  Percentage of Duffy null infants with ANC <1000/µL based on routine CBC performed at at 9-12 months
Association between parental ethnicity and Duffy null phenotype | At birth
  Distribution of Duffy null phenotype stratified by self-reported parental origin.

CONTACTS AND LOCATIONS:
Overall Officials: Tal Ben Ami, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel, Israel

IPD SHARING:
Plan to Share IPD: No
The study involves neonates and is based on anonymized samples; individual-level data will not be shared due to privacy and ethical considerations.

REFERENCES:
- [Background] Gay K, Dulay K, Ravindranath Y, Savasan S. Duffy-Null Phenotype-Associated Neutropenia is the Most Common Etiology for Leukopenia/Neutropenia Referrals to a Tertiary Children's Hospital. J Pediatr. 2023 Nov;262:113608. doi: 10.1016/j.jpeds.2023.113608. Epub 2023 Jul 6. PMID 37419240
- [Background] Rappoport N, Simon AJ, Lev A, Yacobi M, Kaplinsky C, Weingarten M, Somech R, Amariglio N, Rechavi G. Correlation between 'ACKR1/DARC null' polymorphism and benign neutropenia in Yemenite Jews. Br J Haematol. 2015 Sep;170(6):892-5. doi: 10.1111/bjh.13345. Epub 2015 Mar 26. No abstract available. PMID 25817587
- [Background] Atallah-Yunes SA, Ready A, Newburger PE. Benign ethnic neutropenia. Blood Rev. 2019 Sep;37:100586. doi: 10.1016/j.blre.2019.06.003. Epub 2019 Jun 21. PMID 31255364